CLINICAL TRIAL: NCT06301217
Title: Are Axioscapular Muscles Activity and Cervical Curvature Associated With Disability in Patients With Chronic Nonspecific Neck Pain? - A Cross Sectional Exploratory Study
Brief Title: Are Axioscapular Muscles Activity and Cervical Curvature Associated With Disability in Neck Pain
Status: Active, not recruiting | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Omar Mohamed Ali Elabd, Lecturer of Orthopedic Physical Tehrapy, Delta University for Science and Technology
Other Study IDs: NO: PT. BU. EC. 7
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Neck Pain; Electromyohgraph
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: There is no intervention — There is no intervention

SUMMARY:
Despite the important role of axioscapular muscles electromyography and cervical posture as outcomes for the management of chronic neck non specific pain , there is gab of evidence that highlight their association to the commonly used neck disability index. The quest to improve outcomes for individuals suffering from chronic nonspecific neck pain is underscored by the need to identify key prognostic variables that can guide clinical decision-making and intervention strategies. This study seeks to bridge the gap in research by examining the association between neck disability index score, cervical sagittal curvature, and axioscapular muscles electromyography in forms of both trapezius and levator scapula root mean squares to indicate muscular activities and median frequencies to indicate muscular fatigue.

ELIGIBILITY:
Inclusion Criteria:

* chronic nonspecific neck pain
* age between 20 and 40 years,
* either sex
* symptoms lasting longer than three months

Exclusion Criteria:

* Pregnancy
* Spinal surgeries
* spinal deformities
* visual or auditory issues
* ongoing physical or medical treatment for cervical or low back pain

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with chronic nonspecific neck pain lasting longer than three months
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-12-17 (Actual); Primary Completion 2024-03-10 (Estimated); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
Neck disability | at the enrollment
  Neck disability will be measured using the neck disability index. It is a 10-item questionnaire. The patient will be asked to respond by selecting the checkbox next to each statement that most accurately reflect him/her.
Curvature angle of the cervical spine | at the enrollment
  A flexible ruler (ati, FC-700R, Taiwan) will be used to measure the cervical spine curve. To calculate the angle, the patient's elbows will be resting on the armrest directly below the acromion as the patient sat in a chair with his feet flat on the floor, and the ruler will firmly press against the patient's upright cervical spine between the occiput and the seventh cervical spinous process. A mathematical equation will be used: angle (Q)
  =arc tan (2b / a). whereas: a, Length between the two endpoints of the cervical curve; b, Length of the perpendicular from the midpoint of line a to the curve
root-mean-square value (RMS) of Surface electromyography for both upper trapezius and levator scapula | at the enrollment
  electromyography (MyoSystemTM 1400A, Noraxon Inc, 15770 N) will be used to measure:
  * the maximum voluntary isometric contraction of both upper trapezius and levator scapula for 3 trials.
  * Writing task electromyography amplitude for 15 minutes, a semistatic load, after the MVIC evaluation
  Finally, root-mean-square value (%) of both upper trapezius and levator scapula will be calculated as : Writing task electromyography amplitude divided by the average of the three maximum voluntary isometric contraction trials.

CONTACTS AND LOCATIONS:
Locations (1):
- Delta university for science and technology, Gamasa, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Personal preference